CLINICAL TRIAL: NCT07023588
Title: A Multicenter, Open-label, Prospective, Randomized Controlled Study to Optimize the Treatment of Patients With Acute Myeloid Leukemia Based on Early Peripheral Blood Minimal Residual Disease
Brief Title: Study on Optimizing the Treatment of Patients With Acute Myeloid Leukemia Based on Early Peripheral Blood Minimal Residual Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yehui Tan (Other)
Responsible Party: Sponsor-Investigator, Yehui Tan, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-HS-002
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- venetoclax，8-14d (Experimental)
  Interventions: Drug: Venetoclax
- Control group (No Intervention)

INTERVENTIONS:
Drug: Venetoclax — Patients identified with a suboptimal response to chemotherapy based on minimal residual disease (MRD) levels in peripheral blood on Day 6 will initiate venetoclax therapy added on Day 8, administered for 7 days.
  Arms: venetoclax，8-14d

SUMMARY:
A multicenter, open-label, prospective, randomized controlled study to optimize the treatment of patients with acute myeloid leukemia based on early peripheral blood minimal residual disease

DETAILED DESCRIPTION:
This study is a randomized controlled, prospective clinical trial, with the leading unit being the First Hospital of Jilin University. It aims to screen patients with a suboptimal response to chemotherapy based on early peripheral blood minimal residual disease (MRD) levels, and explore the efficacy and safety of adding venetoclax. A total of 70 subjects are expected to be enrolled, with 35 subjects each in the experimental group and the control group. The study will collect data on subjects' demographics, other baseline characteristics, medication usage, prognosis, etc. Statistical analysis will be performed on the collected data to compare efficacy indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML patients confirmed by bone marrow morphology and immunophenotyping.
2. Complete MICM (Morphology, Immunophenotyping, Cytogenetics, Molecular genetics) work-up.
3. Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Day 6 Peripheral Blood Blast Percentage (D6PBBP) ≥ 1%.
6. Renal function with creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula or measured by 24-hour urine collection).
7. Liver function with Aspartate Aminotransferase (AST) ≤ 2.5 × ULN*; Alanine Aminotransferase (ALT) ≤ 2.5 × ULN*; Total bilirubin ≤ 1.5 × ULN* (*Unless considered due to leukemia infiltration).
8. Patients deemed suitable to receive DA/IA therapy by the investigator.
9. Signed informed consent form. -

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL).
2. Mixed phenotype acute leukemia (MPAL).
3. AML patients with known central nervous system (CNS) involvement.
4. Presence of extramedullary disease (EMD).
5. Significant hepatic or renal dysfunction exceeding the inclusion criteria limits.
6. Severe cardiac disease, including congestive heart failure, myocardial infarction, or cardiac dysfunction.
7. Concurrent active malignancy of other organ systems (patients with a history of cured malignancy may be eligible).
8. Active tuberculosis or HIV-positive patients.
9. Concurrent other hematological disorders.
10. Pregnant or lactating women.
11. Inability to comprehend or comply with the study protocol.
12. Hypersensitivity to any component of the drugs involved in the protocol.
13. Inability to take oral medication or patients with malabsorption syndrome.
14. Uncontrolled systemic infection.
15. Prior venetoclax treatment and/or current participation in any other study involving investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Modified Composite Complete Response Rate（mCRc） | Through study completion, an average of 1 year
  Complete Response（CR） + Complete Response with Incomplete Hematologic Recovery（CRi）+Morphologic Leukemia Free State（MLFS）

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 48 months.
  Defined as the time from enrollment in this study to death from any cause. If the exact date of death is unknown, the time of death is defined as the last contact date. If the patient is still alive, the last observed time will be used, and the patient's OS will be considered for analysis.
MRD Negative Conversion Rate | Through study completion, an average of 1 year
  Defined as the proportion of patients who convert to MRD negative among all evaluable patients for efficacy.
Relapse-Free Survival(RFS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 48 months.
  Defined as the time from enrollment in this study to the occurrence of relapse. For patients without relapse, the time is calculated until death from any cause or the time of the last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China